CLINICAL TRIAL: NCT04127617
Title: Neurogenic Bowel Dysfunction: Evaluation of the Effects of Osteopathic Manipulative Treatment in People With Central Nervous System Injury
Brief Title: Effects of Osteopathic Manipulative Treatment in People With Neurogenic Bowel Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: SOMA Istituto Osteopatia Milano (Unknown); A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Alessio Conti, RN, PhD - Postoctoral Fellow in Nursing, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0040534
Record Dates: First submitted 2019-10-04; First posted 2019-10-15 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Central Nervous System Injury; Neurogenic Bowel Dysfunction
Keywords: Manipulation, Osteopathic; Neurogenic Bowel; Nervous System Diseases; Nursing
MeSH Terms: conditions — Neurogenic Bowel; Nervous System Diseases | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. Participants in the study will be divided into two groups: the treatment group will receive five osteopathic manipulative treatment sessions in addition to the standard treatment, and the control group will only receive standard treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): the treatment group will receive 5 osteopathic manipulative treatment. The treatment will last 45 - 60 minutes with the following frequency: the subjects will receive 3 OMT on a weekly basis, the two following twice weekly. The osteopathic treatment protocol will therefore last 7 weeks. Each individual patient will be taken in charge by two operators during the entire duration of the study.
  Interventions: Other: Osteopathic Manipulative Treatment; Other: Nursing Educational Care
- Nursing Care (Active Comparator): The conventional treatment consists in educational nursing care.
  Interventions: Other: Nursing Educational Care

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — Osteopathic treatment
  Dural system:
  L5-S1 decompression; sacred decompression among the iliacs; occipital-sphenoid approach; decongestion of occipital condyles
  Fascial system:
  fascial techniques in the abdominal region: right hypochondrium, epigastrium, left hypochondrium, right side, mesogastrium, left side, right iliac area, hypogastrium, left iliac area; relationship with corresponding vertebral levels (eg, hypogastrium); fibro scar adhesions treatment.
  Biomechanical system:
  diaphragm rebalancing with respect to anatomical insertions; passive mobilization of dysfunctional areas. Nursing education as described in Standard Treatment
  Other Names: Experimental treatment combining osteopathic manipulative treatment with nursing education
  Arms: Osteopathic Manipulative Treatment
Other: Nursing Educational Care — Nursing education
  * assessment of the best personal evacuation strategy concerning the quality of life, individual resources, and level of autonomy;
  * assessment of the correct execution of the identified evacuation manoeuvre (digital stimulation, manual removal, reflex stimulation, transanal irrigation, use of micro-enemas or suppositories;
  * identification of the best postural strategies during evacuation;
  * nutrition and proper hydration education;
  * education in completing the evacuation diary;
  * colonic massage training;
  * verification of the correct hiring of any previously prescribed laxative drugs.
  Other Names: Standard Treatment

SUMMARY:
People affected central nervous system (CNS) diseases often suffer from neurogenic bowel dysfunction (NBD) that causes a reduction in the quality of life and participation in social life. Although some conservative approaches exist to treat NBD, none has shown to be effective in managing this complex condition. Osteopathic manipulative treatment (OMT) has shown to be efficient in CNS diseases such as epilepsy and migraine.

This randomised trial aims at evaluating the efficacy of osteopathic manipulative treatment (OMT) in supporting the management of NBD. The research will be conducted at the outpatient service of Neuro-Urology / Spinal Unit of the Città della Salute e della Scienza Hospital of Torino.

A sample of 62 participants will be divided into two groups: standard (nursing intervention) and experimental (nursing intervention and OMT). A neuro-urologist will determine the eligibility for the study. The outcomes will include self-reported and instrumental measures that will be evaluated in 3 times (before, at the end of the intervention and the follow- up three months).

The protocol has been approved by the Ethics Committee of the Città della Salute e della Scienza Hospital of Torino on 15.04.2019, protocol number 0040534. The standard intervention has been scheduled for 28.10.2019.

DETAILED DESCRIPTION:
Aim of the study The present randomised trial aims to evaluate the efficacy of osteopathic manipulative treatment in supporting the management of neurogenic bowel dysfunction in CNS diseases.

Study design Randomised controlled trial. Participants recruited will be divided into two groups. The treatment group will receive five osteopathic manipulative treatment sessions in addition to the standard treatment.

The control group will only receive standard treatment.

Sample A neuro-urologist will determine eligibility for the study during an interview. Participants will be conducted during outpatient visits to the Neuro Urology department. This study does not include any diagnostic assessment or treatment, which are different from the normal patient's evaluation and management process.

Informed consent will be obtained before any evaluation or treatment. Principal Investigator will explain in detail the study purpose and procedures, risks and potential benefits. Participants will be provided with contact information and have adequate time to consider their participation in the study and encouraged to ask questions, both during the initial interview and throughout the study.

Staff involved in the study Operative Unit Staff (1 urologist specialist, 1 nursing coordinator, 2 nurses); Osteopaths of the School of Osteopathy of Milan (SOMA) who administer osteopathic manipulative treatment; Researcher performing randomisation and data analysis.

Interventions

Eligible participants will be randomised in two different treatment groups:

Conventional therapy (control group)

The conventional treatment consists of education provided by qualified nurses through an individual interview of 45-60 minutes structured as follows:

assessment of the best personal evacuation strategy concerning the quality of life, resources, and level of autonomy; evaluation of the correct execution of the identified evacuation manoeuvre (digital stimulation, manual removal, reflex stimulation, transanal irrigation, use of micro-enemas or suppositories; identification of the best postural strategies during an evacuation; nutrition and proper hydration education; education in completing the evacuation diary; bowel massage training; verification of the correct hiring of any previously prescribed laxative drugs. Approximately two months later, patients will be contacted by telephone to assess the effectiveness of the strategies used to carry out any telephone nursing counselling.

Osteopathic manipulative treatment (experimental group)

In addition to the conventional treatment described above, the experimental group will receive osteopathic manipulative treatment (OMT).

The treatment will last 45 - 60 minutes with the following frequency: the subjects will receive three OMT every week, the two following twice weekly. The osteopathic treatment protocol will, therefore, last seven weeks. Each patient will be taken in charge by two operators during the entire duration of the study.

OMT procedures will be provided by a team of osteopaths, who will practice through specific training to improve palpation reliability before enrollment. The diagnostic and treatment procedures will follow a specific protocol, developed from clinical experience and evidence to improve treatment specificity, safety and reproducibility.

Osteopathic assessment General assessment: the presence of asymmetries, scars. The observation can provide a lot of information on the fascial structure; Assessment of the dural system: cranial and sacral grip, evaluating its intrinsic motility;

Assessment of the fascial system:

lower extremity intrarotation tests and upper limb flexion tests, assesses their quality and amount of movement and any restrictions; abdominal palpation, fascial entrainment in the abdominal-pelvic region; thoracic palpation, fascial entrainment in thoraco-abdominal area.

Assessment of the biomechanical system:

Diaphragms: pelvic, respiratory, upper thoracic, cranial; Structural palpation, spring test: iliac crests, hip mobility, ribs, glenohumeral / clavicles, supine vertebral test.

Each level of assessment (fascial, dural or biomechanical) in which dysfunction is highlighted will be correlated with all other systems and with autonomous nervous system. In relation to the dysfunctions found in the various systems, using parameters such as alterations of tissue density, asymmetry, rigidity (or reduction of range of motion) and tenderness (TART), treatment procedures will be implemented in the specific subject areas at somatic dysfunction.

Osteopathic treatment

Dural system:

L5-S1 decompression; sacred decompression among the iliacs; occipital-sphenoid approach; decongestion of occipital condyles

Fascial system:

fascial techniques in the abdominal region: right hypochondrium, epigastrium, left hypochondrium, right side, mesogastrium, left side, right iliac area, hypogastrium, left iliac area; relationship with corresponding vertebral levels (e.g. hypogastrium); fibro scar adhesions treatment.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic bowel dysfunction secondary to acquired disease of the central nervous system
* Neurogenic Bowel Dysfunction Score (NBDS) between 6 and 30

Exclusion Criteria:

* previous dysfunctional conditions or organic diseases affecting the bowel tract that are pre-existing at neurological diagnosis
* patients with an NBDS score lower than 6 (very mild bowel dysfunction) and above 30 (very severe neurogenic bowel dysfunction)
* ostomy condition (ileus and colon)
* psychiatric patients
* presence of cognitive disorders
* female patients with proven, or even doubtful, pregnancy status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-28 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Neurogenic bowel dysfunction score (NBDS) | - Pre-treatment - Immediately after the treatment - Follow-up at three months after the end of the treatment
  self-reported questionnaire. The Neurogenic Bowel Dysfunction Score is a 10-item questionnaire covering frequency of bowel movements, headache, perspiration or discomfort during defaecation; medication for constipation or faecal incontinence; time spent on defaecation; frequency of digital stimulation or evacuation; frequency of faecal incontinence; flatus; and perianal skin problems. It ranges between 0 and 47; lower scores indicate a better bowel function, while a score over 14 is considered to be an index of severe bowel dysfunction.
  Score 0-6 Very low 7-9 Low 10-13 Moderate 14 or more Severe The hypothesis of treatment efficacy is supported by the observation of a difference between the groups in the NBDS score.

SECONDARY OUTCOMES:
Quality of Life Short Form-36 (SF-36) Questionnaire | - Pre-treatment - Immediately after the treatment - Follow-up at three months after the end of the treatment
  self-reported questionnaire. This questionnaire was developed in 1992 to be applied in all health conditions and detect fundamental human values that describe health concepts significant to a person's functional status and wellbeing. It consists of 36 self-administered questions covering eight main domains (vitality, physical functioning, bodily pain, general health, physical role functioning, emotional role functioning, social role functioning, and mental health) represented on a 0-100 scale; a lower score indicates lower quality of life with significant impairments in the specific domain. Higher scores indicate better quality of life in the different domains.
Bowel transit time | - Pre-treatment - Follow-up at three months after the end of the treatment
  Bowel transit time is a non - invasive diagnostic rx. The exam involves the assumption of radiopaque markers of about two or three millimeters each for six consecutive days and the execution of a single radiograph of the abdomen on the seventh day.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Manassero, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- Silvia Mozzone, Vezza d'Alba, CN, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coggrave M, Norton C, Cody JD. Management of faecal incontinence and constipation in adults with central neurological diseases. Cochrane Database Syst Rev. 2014 Jan 13;2014(1):CD002115. doi: 10.1002/14651858.CD002115.pub5. PMID 24420006
- [Background] Faaborg PM, Christensen P, Buntzen S, Laurberg S, Krogh K. Anorectal function after long-term transanal colonic irrigation. Colorectal Dis. 2010 Oct;12(10 Online):e314-9. doi: 10.1111/j.1463-1318.2010.02198.x. PMID 20070334
- [Background] Gstaltner K, Rosen H, Hufgard J, Mark R, Schrei K. Sacral nerve stimulation as an option for the treatment of faecal incontinence in patients suffering from cauda equina syndrome. Spinal Cord. 2008 Sep;46(9):644-7. doi: 10.1038/sc.2008.6. Epub 2008 Mar 4. PMID 18317481
- [Background] Lombardi G, Del Popolo G, Cecconi F, Surrenti E, Macchiarella A. Clinical outcome of sacral neuromodulation in incomplete spinal cord-injured patients suffering from neurogenic bowel dysfunctions. Spinal Cord. 2010 Feb;48(2):154-9. doi: 10.1038/sc.2009.101. Epub 2009 Aug 11. PMID 19668257
- [Background] Schleip R, Muller DG. Training principles for fascial connective tissues: scientific foundation and suggested practical applications. J Bodyw Mov Ther. 2013 Jan;17(1):103-15. doi: 10.1016/j.jbmt.2012.06.007. Epub 2012 Jul 21. PMID 23294691
- [Background] Branchini M, Lopopolo F, Andreoli E, Loreti I, Marchand AM, Stecco A. Fascial Manipulation(R) for chronic aspecific low back pain: a single blinded randomized controlled trial. F1000Res. 2015 Nov 3;4:1208. doi: 10.12688/f1000research.6890.2. eCollection 2015. PMID 26834998
- [Background] Ruffini N, D'Alessandro G, Mariani N, Pollastrelli A, Cardinali L, Cerritelli F. Variations of high frequency parameter of heart rate variability following osteopathic manipulative treatment in healthy subjects compared to control group and sham therapy: randomized controlled trial. Front Neurosci. 2015 Aug 4;9:272. doi: 10.3389/fnins.2015.00272. eCollection 2015. PMID 26300719
- [Background] Tesarz J, Hoheisel U, Wiedenhofer B, Mense S. Sensory innervation of the thoracolumbar fascia in rats and humans. Neuroscience. 2011 Oct 27;194:302-8. doi: 10.1016/j.neuroscience.2011.07.066. Epub 2011 Aug 2. PMID 21839150
- [Background] Licciardone JC, Kearns CM, Hodge LM, Bergamini MV. Associations of cytokine concentrations with key osteopathic lesions and clinical outcomes in patients with nonspecific chronic low back pain: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Sep;112(9):596-605. doi: 10.7556/jaoa.2012.112.9.596. PMID 22984233
- [Background] Bramati-Castellarin I, Patel VB, Drysdale IP. Repeat-measures longitudinal study evaluating behavioural and gastrointestinal symptoms in children with autism before, during and after visceral osteopathic technique (VOT). J Bodyw Mov Ther. 2016 Jul;20(3):461-70. doi: 10.1016/j.jbmt.2016.01.001. Epub 2016 Jan 14. PMID 27634066
- See also: International Classification of Disease 10, (2016). Segmental and somatic dysfunction. — http://apps.who.int/classifications/icd10/browse/2016